CLINICAL TRIAL: NCT05013957
Title: Neuroendocrine Neoplasms Methylation Based Classifier - The NEMESIs-study
Acronym: NEMESIs
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: NEMESIs study
Record Dates: First submitted 2021-08-17; First posted 2021-08-20 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Neuroendocrine Tumors
Keywords: Methyloma
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective analysis: Methylome of existing neuroendocrine tumor samples from the biobank of Basel University Hospital will be evaluated
  Interventions: Diagnostic Test: Methylation analysis
- Prospective analysis: Methylome analysis of tumor samples of neuroendocrine tumor patients undergoing an operation or biopsy will be prospectively evaluated
  Interventions: Diagnostic Test: Methylation analysis

INTERVENTIONS:
Diagnostic Test: Methylation analysis — Methylation analysis

SUMMARY:
Neuroendocrine neoplasms (NEN) are rare tumors that mainly occur in the gastrointestinal tract and the lungs. The currently available diagnostic and prognostic markers do not adequately represent the diversity of these tumors. Methylation analyzes of the tumor DNA represent a new, promising approach.

The aim of this project is therefore to improve the diagnostic and prognostic evaluation of neuroendocrine neoplasms by means of methylation analysis of the tumor DNA. On the one hand, existing tumor samples from the biobank of Basel University Hospital are evaluated, on the other hand, patients who are undergoing an operation will be prospectively inquired

ELIGIBILITY:
Inclusion Criteria:

* neuroendocrine tumor

Exclusion Criteria:

* insufficient amount or quality of neuroendocrine tumor sample

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neuorendocrine tumor patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Methylation-based classification of NEN samples | 3 years
  NEN samples will be classified according to methylation analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Department of Endocrinology, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided